CLINICAL TRIAL: NCT04040634
Title: Large-Scale Randomized Clinical Trial Assessing Intensive Blood Pressure Control for Reduction of Major Cardiovascular Events in Patients With Diabetes Mellitus (OPTIMAL-DIABETES)
Brief Title: Optimal Blood Pressure for the prevenTIon of Major vAscuLar Events in Patients With DIABETES Mellitus (OPTIMAL-DIABETES)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Israelita Albert Einstein (Other)
Collaborators: Ministry of Health, Brazil (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OPTIMAL-DIABETES Trial; 02795218.8.1001.0071 (Other: Plataforma Brasil (CAAE #)); 25000.028978/2018-02 (Other Grant/Funding Number: Ministry of Health, Brazil (NUP#))
Record Dates: First submitted 2019-07-30; First posted 2019-08-01 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-10

CONDITIONS: Diabetes Mellitus; High Blood Pressure; Cardiovascular Diseases; Cognitive Impairment
MeSH Terms: conditions — Diabetes Mellitus; Hypertension; Cardiovascular Diseases; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensive Control of Systolic Blood Pressure (SBP) (Experimental): Participants randomized into the Intensive Blood Pressure arm will have a goal of SBP <120 mm Hg.
  Interventions: Drug: Intensive Control of Systolic Blood Pressure (SBP)
- Standard Control of Systolic Blood Pressure (SBP) (Active Comparator): Participants randomized into the Standard arm will have a goal of SBP <140 mm Hg.
  Interventions: Drug: Standard control of Systolic Blood Pressure (SBP)

INTERVENTIONS:
Drug: Intensive Control of Systolic Blood Pressure (SBP) — Participants in the Intensive arm have a goal of SBP <120 mm Hg. The use of angiotensin converting enzyme (ACE) inhibitors/angiotension receptor blockers (ARB), thiazide-type diuretics, and calcium channel blockers (CCB) will be encouraged, preferably fixed-dose combinations of indapamide + perindopril arginine, perindopril arginine + amlodipine or indapamide + perindopril arginine + amlodipine
  Other Names: Intensive BP control targeting SBP <120 mm Hg
  Arms: Intensive Control of Systolic Blood Pressure (SBP)
Drug: Standard control of Systolic Blood Pressure (SBP) — The same medications used in the Intensive BP arm will be used for the Standard BP arm.
  Other Names: Standard control of SBP targeting SBP < 140 mm Hg
  Arms: Standard Control of Systolic Blood Pressure (SBP)

SUMMARY:
High blood pressure (BP) is a major public health concern, especially in low and middle income countries. High BP is a highly prevalent condition, and it is usually associated with diabetes mellitus. Both high BP and diabetes are risk factors for major cardiovascular events including cardiovascular death, acute myocardial infarction, stroke, unstable angina and heart failure. In addition, high BP is also related to cognitive decline. The OPTIMAL-DIABETES trial consists of a two-arm, multicenter, randomized clinical trial designed to test whether a lower systolic blood pressure (SBP) target will reduce the occurrence of major cardiovascular events in diabetic patients compared to the standard SBP target.

ELIGIBILITY:
Inclusion Criteria:

* Systolic Blood Pressure (SBP) between 130 and 180 mm Hg:

  * 130 to 150 mm Hg (if on 0-4 medications)
  * 130 to 160 mm Hg (if on 0-3 medications)
  * 130 to 170 mm Hg (if on 0-2 medications)
  * 130 to 180 mm Hg (if on 0-1 medications)
* Type 2 diabetes
* To be considered as having a high cardiovascular risk, including AT LEAST ONE of the following factors:

  1. Established cardiovascular disease (CVD), including:

     * Coronary artery disease: previous myocardial infarction, previous acute coronary syndrome, previous percutaneous coronary intervention, previous coronary artery bypass graft surgery, or at least 50% stenosis in a main coronary artery associated with typical angina pectoris; or
     * Cerebrovascular disease: previous stroke (except those events caused by intracranial aneurysm or arteriovenous malformation) or previous transient ischemic attack (TIA), stable for at least 2 weeks preceding inclusion in the study; or
     * Carotid artery disease: previous carotid endarterectomy, previous percutaneous intervention with carotid stent implantation, or stenosis of at least 50% in a carotid shown by the Doppler ultrasonography, CT angiography or MR angiography; or
     * Peripheral artery disease: prior surgical or percutaneous revascularization of a peripheral artery, limb amputation due to vascular cause, abdominal aortic aneurysm ≥ 5 cm (with or without prior surgical or percutaneous repair), or stenosis of at least 50% in a peripheral artery associated to intermittent claudication.
  2. Subclinical CVD, including:

     * Coronary calcium score ≥ 300 Agatston units; or
     * Ankle-brachial index ≤ 0.90 in the last two years; or
     * Left ventricular hypertrophy on the electrocardiogram, echocardiogram or other cardiac imaging exam in the last two years.
  3. Chronic kidney disease (CKD):

     ▪ Definition of CKD: glomerular filtration rate (GFR) between 20 and 59 ml/min/1.73m2 calculated by the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI).
  4. Additional cardiovascular risk factors, including:

     * Active smoking: Defined as regular use of cigarettes or other tobacco products, such as cigars and pipe, in the last six months;
     * Dyslipidemia: Defined as LDL cholesterol > 70 mg/dL or non-HDL cholesterol > 100 mg/dL in patients with previous CVD; or LDL cholesterol > 100 mg/dL or non-HDL cholesterol > 130 mg/dL in patients without previous CVD; or Triglycerides > 200 mg/dL or HDL < 40 mg/dL regardless of treatment; or use of statins or other lipid lowering medication; or
     * Age ≥ 75 years

Exclusion Criteria:

* Refusal to provide written informed consent
* Body mass index > 45 kg/m2
* Known secondary cause of hypertension
* Severe renal dysfunction with GFR < 20 mL/min/1.73m2 calculated by the CKD-EPI equation
* Angina at rest Class IV Canadian Cardiovascular Society (CCS)
* Acute coronary syndrome in the last six months
* Symptomatic heart failure Class IV New York Heart Association (NYHA) or ejection fraction < 35% on Doppler echocardiography in the last six months
* Factors that at the research team´s judgment may limit adherence to the intervention and study protocol, including, but not limited to, the following examples:

  * Recent history of alcohol and illicit drug abuse
  * Psychiatric comorbidities (severe depression, schizophrenia, psychosis, etc.)
  * History of poor medication adherence and attendance to consultations
  * Any plans to move the city of residence in the next four years
  * Any plans to leave the city of residence for more than three months in the next few years
  * Living in the same residence of another patient previously included in this study
* Patients currently enrolled in another study for CVD prevention, including those evaluating pharmacological and non-pharmacological interventions
* Pregnancy or breastfeeding

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9479 (Actual)
Dates: Start 2019-08-08 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Time to cardiovascular death, non-fatal myocardial infarction (MI), non-fatal stroke, hospitalization for unstable angina or hospitalization for heart failure | From randomization to 48 months
  Time to first event of cardiovascular death, non-fatal myocardial infarction (MI), non-fatal stroke, hospitalization for unstable angina or hospitalization for heart failure

SECONDARY OUTCOMES:
Time to cardiovascular death, non-fatal myocardial infarction (MI) or non-fatal stroke | From randomization to 48 months
  Time to first event of cardiovascular death, non-fatal myocardial infarction (MI) or non-fatal stroke
Time to total death, non-fatal myocardial infarction (MI), non-fatal stroke, hospitalization for unstable angina or hospitalization for heart failure | From randomization to 48 months
  Time to first event of total death, non-fatal myocardial infarction (MI), non-fatal stroke, hospitalization for unstable angina or hospitalization for heart failure
Time to Death | From randomization to 48 months
  Time to all cause death
Time to Cardiovascular Death | From randomization to 48 months
  Time to death from cardiovascular causes
Time to Renal Death | From randomization to 48 months
  Time to death from renal causes
Time to Myocardial Infarction (MI) | From randomization to 48 months
  Time to myocardial infarction (MI)
Time to Stroke | From randomization to 48 months
  Time to stroke
Time to Ischemic Stroke | Follow-up of 48 months
  Time to ischemic stroke
Time to Hemorrhagic Stroke | From randomization to 48 months
  Time to hemorrhagic stroke
Time to Undetermined type of Stroke | From randomization to 48 months
  Time to Undetermined type of Stroke
Time to Transient Ischemic Attack (TIA) | From randomization to 48 months
  Time to transient ischemic attack (TIA)
Time to Hospitalization for Unstable Angina | From randomization to 48 months
  Time to Hospitalization for unstable angina
Time to Hospitalization for Heart Failure | From randomization to 48 months
  Time to hospitalization for heart failure
Time to Renal Outcome | From randomization to 48 months
  Time to Renal Outcome, defined as a ≥50% reduction in the glomerular filtration rate (GFR) from baseline (excluding acute reversible causes) or progression to end-stage renal disease, which is defined as a GFR < 15 mL/min/1.73m² (excluding reversible causes) or the need for dialysis (hemodialysis or peritoneal dialysis for at least 30 days) or kidney transplantation
Time to decrease in the Montreal Cognitive Assessment (MoCA) score | From randomization to 48 months
  Time to decrease in the Montreal Cognitive Assessment (MoCA) score
Time to Mild Cognitive Impairment | From randomization to 48 months
  Time to Mild Cognitive Impairment
Time to Mild Cognitive Impairment or All-Cause Probable Dementia | From randomization to 48 months
  Time to mild cognitive impairment or all-cause probable dementia
Time to All-Cause Probable Dementia | From randomization to 48 months
  Time to all-cause probable dementia

CONTACTS AND LOCATIONS:
Overall Officials: Otavio Berwanger, MD, PhD, Study Director — Hospital Israelita Albert Einstein
Locations (32):
- Brazil (32):
  - Centro de Pesquisas Clínicas Dr Marco Mota, Maceió, Alagoas
  - Instituto de Estudos E Pesquisas Clinicas Do Ceara, Fortaleza, Ceará
  - Hospital Universitário Cassiano Antonio de Moraes, Vitória, Espírito Santo
  - Centro de Pesquisas em Diabetes e Doenças Endocrino-Metabólicas, Fortaleza, Estado de Bahia
  - Hospital Ana Nery, Salvador, Estado de Bahia
  - Instituto Hospital de Base, Brasília, Federal District
  - Universidade Federal de Goiás, Goiânia, Goiás
  - NS Clínica de Diabetes e Endocrinologia Ltda, Goiânia, Goiás
  - Hospital das Clinicas da Universidade Federal de Minas Gerais, Belo Horizonte, Minas Gerais
  - Centro de Pesquisa do Hospital Santa Lúcia, Poços de Caldas, Minas Gerais
  - Medicina Nuclear Alto da XV, Curitiba, Paraná
  - Hospital Universitário João de Barros Barreto - UFPA, Belém, Pará
  - Pronto Socorro Cardiológico de Pernambuco Prof. Luiz Tavares da Silva, Recife, Pernambuco
  - Faculdade de Ciências Médicas - Universidade do Estado do Rio de Janeiro, Rio de Janeiro, Rio de Janeiro
  - Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital São Lucas da PUCRS, Porto Alegre, Rio Grande do Sul
  - Centro de Pesquisa Clínica do Coração, Aracaju, Sergipe
  - Centro de Endocrinologia Geloneze, Campinas, São Paulo
  - Universidade Estadual de Campinas - UNICAMP, Campinas, São Paulo
  - Indacor Servicos Medicos Ltda, Indaiatuba, São Paulo
  - Hospital das Clinicas da Faculdade de Medicina de Ribeirão Preto da Universidade de São Paulo, Ribeirão Preto, São Paulo
  - Centro Integrado de Pesquisas, São José do Rio Preto, São Paulo
  - Clínica Vilela & Martin, São José do Rio Preto, São Paulo
  - Instituto de Cardiologia e Endocrinologia Rio Preto Ltda, São José do Rio Preto, São Paulo
  - Clínica de Metabologia e Hipertensão da Universidade Federal de São Paulo, São Paulo, São Paulo
  - Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo, São Paulo
  - Instituto do Coração do Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo, São Paulo
  - Instituto Dante Pazzanese de Cardiologia, São Paulo, São Paulo
  - Irmandade Da Santa Casa de Misericordia de Sao Paulo, São Paulo, São Paulo
  - Real e Benemérita Associação Portuguesa de Beneficência/SP, São Paulo, São Paulo
  - Clínica Cardiológica, Votuporanga, São Paulo
  - Santa Casa de Misericordia de Votuporanga, Votuporanga, São Paulo

REFERENCES:
- [Derived] Saiz LC, Gorricho J, Garjon J, Celaya MC, Erviti J, Leache L. Blood pressure targets for the treatment of people with hypertension and cardiovascular disease. Cochrane Database Syst Rev. 2022 Nov 18;11(11):CD010315. doi: 10.1002/14651858.CD010315.pub5. PMID 36398903
- [Derived] Saiz LC, Gorricho J, Garjon J, Celaya MC, Erviti J, Leache L. Blood pressure targets for the treatment of people with hypertension and cardiovascular disease. Cochrane Database Syst Rev. 2020 Sep 9;9(9):CD010315. doi: 10.1002/14651858.CD010315.pub4. PMID 32905623